CLINICAL TRIAL: NCT05976555
Title: Phase I Study of BCMA-TGF-BETA Insensitive Armored CAR T Cells in Patients With Relapsed and/or Refractory Multiple Myeloma
Brief Title: Phase I Trial of BCMA-TGF-BETA CAR-T Cells in Relapsed, Refractory Myeloma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Binod Dhakal, Associate Professor, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IIT-DHAKAL-TGF-BETA-BCMA
Record Dates: First submitted 2023-07-28; First posted 2023-08-04 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Multiple Myeloma
Keywords: CAR-T; Chimeric antigen receptor T-cell therapy; CAR Therapy
MeSH Terms: conditions — Multiple Myeloma | interventions — Maximum Tolerated Dose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- BCMA-TGFβ CAR-T cells (0.50 x 10^6 cells/kg) (Experimental): BCMA-TGFβ CAR-T cells will be administered either fresh or thawed after cryopreservation by IV injection. Subjects will receive one of four dose levels of BCMA-TGFβ CAR-T cells based on the dose escalation design.
  Interventions: Biological: BCMA-TGFβ CAR-T cells (0.50 x 10^6 cells/kg)
- BCMA-TGFβ CAR-T cells (0.75 x10^6 cells/kg) (Experimental): BCMA-TGFβ CAR-T cells will be administered either fresh or thawed after cryopreservation by IV injection. Subjects will receive one of four dose levels of BCMA-TGFβ CAR-T cells based on the dose escalation design.
  Interventions: Biological: BCMA-TGFβ CAR-T cells (0.75 x10^6 cells/kg)
- BCMA-TGFβ CAR-T cells (1 x 10^6 cells/kg) (Experimental): BCMA-TGFβ CAR-T cells will be administered either fresh or thawed after cryopreservation by IV injection. Subjects will receive one of four dose levels of BCMA-TGFβ CAR-T cells based on the dose escalation design.
  Interventions: Biological: BCMA-TGFβ CAR-T cells (1 x 10^6 cells/kg)
- BCMA-TGFβ CAR-T cells (2.5 x 10^6 cells/kg) (Experimental): BCMA-TGFβ CAR-T cells will be administered either fresh or thawed after cryopreservation by IV injection. Subjects will receive one of four dose levels of BCMA-TGFβ CAR-T cells based on the dose escalation design.
  Interventions: Biological: BCMA-TGFβ CAR-T cells (2.5 x 10^6 cells/kg)
- BCMA-TGFβ CAR-T cells (Maximum tolerated dose) (Experimental): After the maximal tolerated dose (MTD) is determined, an additional dose-expansion cohort of up to 9 patients (3 BCMA-naïve and 6 BCMA exposed) may be enrolled at that dose.
  Interventions: Biological: BCMA-TGFβ CAR-T cells (0.50 x 10^6 cells/kg); Biological: BCMA-TGFβ CAR-T cells (0.75 x10^6 cells/kg); Biological: BCMA-TGFβ CAR-T cells (1 x 10^6 cells/kg); Biological: BCMA-TGFβ CAR-T cells (2.5 x 10^6 cells/kg); Biological: Maximum tolerated dose

INTERVENTIONS:
Biological: BCMA-TGFβ CAR-T cells (0.50 x 10^6 cells/kg) — This is dose level 0 (de-escalation).
  Arms: BCMA-TGFβ CAR-T cells (0.50 x 10^6 cells/kg); BCMA-TGFβ CAR-T cells (Maximum tolerated dose)
Biological: BCMA-TGFβ CAR-T cells (0.75 x10^6 cells/kg) — This is dose level 1, the starting dose.
  Arms: BCMA-TGFβ CAR-T cells (0.75 x10^6 cells/kg); BCMA-TGFβ CAR-T cells (Maximum tolerated dose)
Biological: BCMA-TGFβ CAR-T cells (1 x 10^6 cells/kg) — This is dose level 2.
  Arms: BCMA-TGFβ CAR-T cells (1 x 10^6 cells/kg); BCMA-TGFβ CAR-T cells (Maximum tolerated dose)
Biological: BCMA-TGFβ CAR-T cells (2.5 x 10^6 cells/kg) — This is dose level 3.
  Arms: BCMA-TGFβ CAR-T cells (2.5 x 10^6 cells/kg); BCMA-TGFβ CAR-T cells (Maximum tolerated dose)
Biological: Maximum tolerated dose — The maximum tolerated dose is yet to be determined.
  Arms: BCMA-TGFβ CAR-T cells (Maximum tolerated dose)

SUMMARY:
This is a phase I, interventional, single-arm, open-label, dose-finding treatment study designed to evaluate the safety and efficacy of interleukin-7(IL-7) / interleukin-15 (IL-15) manufactured CAR T cells in adult patients with relapsed and/or refractory myeloma that have failed prior therapies.

DETAILED DESCRIPTION:
BCMA-Transforming growth factor-beta (TGFβ) CAR-T cells will be administered either fresh or thawed after cryopreservation by IV injection. Patients will receive one of three dose levels of BCMA-TGFβ CAR-T cells based on our dose escalation design.

After the maximal tolerated dose (MTD) is determined, an additional dose-expansion cohort of up to 9 patients (3 BCMA-naïve and 6 BCMA exposed) may be enrolled at that dose to further describe the safety and preliminary efficacy of that dose.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be aged ≥18 years to 80 years old.
2. Patients must have received three prior lines of therapies, including proteasome inhibitor, immunomodulator and a cluster of differentiation (CD) 38 monoclonal antibody:

   • International Myeloma Working Group (IMWG) criteria defines refractory disease as disease progression on or within 60 days of receiving therapy.
3. Patients must have measurable disease, including at least one or more of the following criteria:

   1. Serum M-protein ≥0.5 g/dl;
   2. Urine M-protein ≥200 mg/24 hrs;
   3. Involved serum light chain ≥100 mg/L with abnormal light chain ratio;
4. Absolute CD 3 count ≥50 mm^3.
5. Karnofsky performance score ≥70.
6. Adequate hepatic function, defined as:

   1. aspartate aminotransferase (AST), alanine transaminase (ALT), and alkaline phosphatase <3x upper limit of normal (ULN);
   2. Serum bilirubin <2.0 mg/dL except for patients with Gilbert's syndrome, who must have serum bilirubin of <3 mg/dL.
7. Absolute neutrophil count (ANC) ≥1,000 with no Granulocyte colony-stimulating factor (G-CSF) within 72 hours or pegylated G-CSF within 10 days.
8. Platelets ≥50,000/µL with no transfusion within 72 hours of eligibility testing.
9. Adequate renal function, defined as creatinine clearance ≥50 mL/min calculated using the Cockroft-Gault formula.
10. Able to provide written informed consent.
11. Agree to practice birth control during the study.
12. Adequate cardiac function as indicated by New York Heart Association (NYHA) classification I or II AND left ventricular ejection fraction of ≥45% (by cardiac echocardiogram (ECHO) or multigated acquisition (MUGA)) and adequate pulmonary function as indicated by room air oxygen saturation of ≥90%.
13. Expected survival >12 weeks.
14. Negative urine or serum pregnancy test in females of childbearing potential at study entry.
15. Meet criteria for regarding fertility and contraception detailed below.
16. No contraindication to central line access.

Phase I Dose-Expansion Cohort A: BCMA Naïve The inclusion criteria for dose-expansion Cohort A are the same as that listed above but are limited to BCMA naïve patients.

Phase I Dose-Expansion Cohort B: BCMA Exposed The inclusion criteria for dose expansion Cohort B are the same as that above but require prior exposure to BCMA directed therapies (e.g., CAR-BCMA, bispecific T/ Natural Killer (NK) cell engagers of BCMA).

Patients with prior antibody drug conjugate, bispecific T and NK cell engager and prior gene-modified cellular immune therapy against BCMA are allowed. Patients must be > 3 months out from therapy and must have achieved stable disease or better with prior BCMA-directed therapy.

Exclusion Criteria:

1. Positive beta- Human chorionic gonadotropin (HCG) in female of child-bearing potential defined as per the Schedule of Events table.
2. Confirmed active human immunodeficiency virus (HIV), Hepatitis B or C infection.
3. History of significant autoimmune disease OR active, uncontrolled autoimmune phenomenon requiring steroid therapy defined as >20 mg of prednisone or equivalent daily.
4. Presence of ≥ Grade 3 non-hematologic toxicities as per CTCAE version 5.0 from any previous treatment unless it is felt to be due to underlying disease.
5. Concurrent use of investigational therapeutic agents or enrollment on another therapeutic clinical trial at any institution. Minimum of 14 days or 5 half-lives of the drug (whichever is shorter) washout prior to apheresis.
6. Refusal to participate in the long-term follow-up protocol.
7. Patients with active central nervous system (CNS) involvement by malignancy on MRI or by lumbar puncture.

   a. Patients with prior CNS disease that has been effectively treated will be eligible providing last treatment was ≥2 weeks before apheresis and a remission documented within 4 weeks of planned CAR T-cell infusion by MRI brain and CSF analysis.
8. Previous recipients of allogeneic hematopoietic stem cell transplantation (AHCT) are excluded if they are <6 months post-transplant, have evidence of active graft-versus-host-disease (GVHD) of any grade, or are currently on immunosuppression.
9. Plasma cell leukemia, Waldenstrom's macroglobulinemia, POEMS syndrome, and AL amyloidosis.
10. Prior treatment with gene therapy or any gene modified cellular therapy (only permitted in cohort B for the dose expansion phase).
11. Prior BCMA-directed therapy (only permitted in cohort B for the dose expansion phase).
12. Cytotoxic chemotherapy, oral chemotherapeutic agents, or antibody-directed treatment within 14 days of apheresis or after apheresis.

    1. Corticosteroids are allowable up until 7 days prior to apheresis and after apheresis for disease control up until the day prior to cell infusion (Day -1).
    2. Radiation is allowed to a single symptomatic site.
13. Patients post solid organ transplant who develop high grade lymphomas or leukemias.
14. Concurrent active malignancy other than basal or squamous cell carcinomas of the skin.
15. Active bacterial, viral, or fungal infection requiring systemic treatment.
16. Patients who have received major surgery 1 week prior to leukapheresis and 3 weeks prior to lymphodepletion.
17. Active malignancy that required therapy in the last 2 years except successfully treated non metastatic basal or squamous cell carcinoma, or prostate carcinoma that does not require therapy. Other similar conditions may be discussed with and permitted by the medical monitor.

Special Criteria Regarding Fertility and Contraception

Female subjects of reproductive potential (women who have reached menarche or women who have not been post-menopausal for at least 24 consecutive months, i.e., who have had menses within the preceding 24 months, or have not undergone a sterilization procedure [hysterectomy or bilateral oophorectomy]) must have a negative serum or urine pregnancy test performed as part of eligibility criteria. Lactating women are eligible for this study but will be asked to not provide breast milk to their child from Day -4 through Day +90 after CAR T-cell therapy.

Due to the high-risk level of this study, while enrolled, all subjects must agree not to participate in a conception process (e.g., active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization). Additionally, if participating in sexual activity that could lead to pregnancy, the study subject must agree to use reliable and double barrier methods of contraception during the follow-up period of the protocol.

Acceptable birth control includes a combination of two of the following methods:

* Condoms (male or female) with or without a spermicidal agent.
* Diaphragm or cervical cap with spermicide.
* Intrauterine device (IUD).
* Hormonal-based contraception. Subjects who are not of reproductive potential (women who are premenarche or have been post-menopausal for at least 24 consecutive months or have undergone hysterectomy, tubal ligation, salpingectomy, and/or bilateral oophorectomy or men who have documented azoospermia) are eligible without requiring the use of contraception.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events After BCMA-TGFβ CAR-T Cell Infusion | from infusion until Day +28 post CAR T infusion
  Incidence of adverse events with grade 3 to 5 severity using NCI CTCAE version 5.0 and the Lee et al. consensus manuscript (which outlines the defining characteristics of each grade for cytokine release syndrome; please refer to the reference below).

CONTACTS AND LOCATIONS:
Overall Officials: Binod Dhakal, MD, Principal Investigator — Medical College of Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee DW, Santomasso BD, Locke FL, Ghobadi A, Turtle CJ, Brudno JN, Maus MV, Park JH, Mead E, Pavletic S, Go WY, Eldjerou L, Gardner RA, Frey N, Curran KJ, Peggs K, Pasquini M, DiPersio JF, van den Brink MRM, Komanduri KV, Grupp SA, Neelapu SS. ASTCT Consensus Grading for Cytokine Release Syndrome and Neurologic Toxicity Associated with Immune Effector Cells. Biol Blood Marrow Transplant. 2019 Apr;25(4):625-638. doi: 10.1016/j.bbmt.2018.12.758. Epub 2018 Dec 25. PMID 30592986